CLINICAL TRIAL: NCT01722968
Title: A Prospective Randomized Phase II Study to Identify Predictive Biomarkers and Mechanisms of Therapy Resistance in Patients With HER2-negative Metastatic Breast Cancer Treated With the Combination of Bevacizumab and Paclitaxel (BEVPAC).
Brief Title: A Biomarker Study in Patients With HER2-negative Metastatic Breast Cancer Treated With Bevacizumab and Paclitaxel
Acronym: BEVPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theodoros Foukakis (Other)
Responsible Party: Sponsor-Investigator, Theodoros Foukakis, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT no: 2012-003743-30
Record Dates: First submitted 2012-10-22; First posted 2012-11-07 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Arm A and feasibility phase: Bevacizumab 15mg/kg administered iv every 3 weeks in combination with paclitaxel 80mg/m2 iv weekly.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel
- Arm B (Active Comparator): Arm B: Paclitaxel 80mg/m2 iv weekly.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — 15mg/kg administered iv every 3 weeks in combination with paclitaxel 80mg/m2 iv weekly
  Other Names: Avastin
  Arms: Arm A
Drug: Paclitaxel — 80mg/m2 iv weekly
  Other Names: Paxene; Taxol

SUMMARY:
To explore molecular biomarkers and/or gene expression signatures that predict response to bevacizumab given in combination with paclitaxel as first line therapy in HER2 negative metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
This is a prospective, randomized, 2-arm, open-label, single-center, phase II trial. A total of 30 patients will be included during a period of 2 years.

The study will be initiated with a non-randomized, feasibility stage including ten patients who will be treated with bevacizumab and paclitaxel, in order to determine the safety of metastatic tumor biopsies during therapy with bevacizumab.

In the second phase, patients will be randomized (1:1) between two treatment arms: A. Bevacizumab + paclitaxel and B. Paclitaxel

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. Performance status ECOG 0-2.
3. Clinically and / or radiologically proven stage IV or recurrent HER2 negative breast cancer.
4. At least one tumor lesion accessible for biopsy. This lesion may not have been treated previously with irradiation.
5. Clinically and/or radiographically documented measurable disease according to RECIST v1.1 criteria. At least one site of disease must be unidimensionally measurable as follows:

   1. CT-scan, physical exam ≥ 10 mm} Chest X-ray ≥ 20 mm }see Eisenhauer et al. for more details
   2. Lymph node short axis ≥ 15 mm }
   3. All radiology studies must be performed within 28 days prior to registration (35 days if negative).
6. Adequate bone-marrow, hepatic and renal function defined as laboratory tests within 7 days prior to enrollment:

   1. Haematology: Absolute granulocytes > 1.5 x 109/L Platelets > 100 x 109/L
   2. Biochemistry:Bilirubin within normal limits Serum creatinine within normal limits
7. APTT and INR within normal limits within 7 days prior to enrollment.
8. Adequate cardiac function with Left Ventricular Ejection Fraction (LVEF) within normal limits determined by echocardiogram or MUGA within 28 days prior to inclusion.
9. Written informed consent must be given.

Exclusion Criteria:

1. Previous systemic treatment for MBC.
2. Major surgery less than 28 days prior to enrollment.
3. Concurrent malignancy of any site, except adequately controlled limited basal cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix.
4. Bleeding diathesis, history of thromboembolic disease, or ongoing treatment with warfarin, heparin analogs or antiplatelet drugs.
5. Major cardiac comorbidity.
6. Previous treatment with bevacizumab.
7. Previous allergic reaction to taxane analogs.
8. Ongoing pregnancy or lactation.
9. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-11; Primary Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Identification of molecular biomarkers | After the study completion,After completion of the study, which will take up to 3 years
  To explore molecular biomarkers and/or gene expression signatures that predict response to bevacizumab given in combination with paclitaxel as first line therapy in HER2 negative MBC.

SECONDARY OUTCOMES:
Safety of metastatic biopsies during bevacizumab therapy | continuous assessment and after inclusion of 10 patients, After completion of the study which will take up to 1 year
  The safety objective of the study is to assess whether carrying out metastatic tissue biopsies during treatment with bevacizumab is safe. For this reason, the study will be initiated with a feasibility phase of 10 patients and will be continued to the randomized phase only if the study specific procedures prove to be safe.

OTHER OUTCOMES:
Molecular changes by bevacizumab | After completion of the study which will take up to 3 years
  To identify molecular changes in the tumor induced by the addition of bevacizumab to chemotherapy.
Efficacy of bevacizumab | After completion of the study, After completion of the study, which will take up to 3 years
  To measure the efficacy of bevacizumab in combination with paclitaxel in HER2 negative MBC.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Foukakis, MD PhD, Principal Investigator — Karolinska University Hospital; Jonas Bergh, Professor, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Solna, Stockholm County, Sweden